CLINICAL TRIAL: NCT06859112
Title: The Effect of Logotherapy-Based Psychoeducation Applied to Family Members of Individuals Diagnosed with Schizophrenia on Finding Meaning, Hope and Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: aslı zeynep sipahi (Other)
Responsible Party: Sponsor-Investigator, aslı zeynep sipahi, lecturer, Uskudar University
Organization: Uskudar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 61351342Ekim/2022 21
Record Dates: First submitted 2024-12-30; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia, psychoeducation, patient's relative, logotherapy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: This research was planned as a mixed design study in which quantitative and qualitative approaches were used together. The quantitative phase of the research consists of a prospective, single-blind, randomized controlled study design using a pre-test-post-test design aiming to reveal the effectiveness of Logotherapy-Based Psychoeducation. The qualitative phase of the study will be applied with a phenomenological approach to clarify the attitude changes of the participants in the experimental group during and after the Logotherapy-Focused Psychoeducation Program.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Relatives of patients who underwent the application (Experimental): Individuals in this group will receive 8 sessions of psychoeducation focused on logotherapy.
  Interventions: Other: logotherapy focused psychoeducation
- relatives of patients in routine practice (No Intervention): Individuals in this arm will not be subjected to any additional intervention other than routine practices.

INTERVENTIONS:
Other: logotherapy focused psychoeducation — 8 sessions of online individual logotherapy focused psychoeducation program
  Arms: Relatives of patients who underwent the application

SUMMARY:
The resources that will strengthen the family members who play a key role in the treatment of schizophrenia should also be activated. One of these resources that enable people to cope with the difficult events they experience is finding meaning in life. The meaning of life is a basic source of motivation for an individual to live despite everything. In this respect, meaning is a source that helps them maintain their mental balance. Another concept that is considered important in terms of protecting and strengthening the mental health of family members is hope. Hope is defined as setting a goal and taking action to achieve it, and looking for different ways when faced with difficulties. Hope gives caregivers the belief that they can cope with stressful experiences. Therefore, it is important to develop hope in family members of individuals with mental disorders. Today, different therapy methods are applied to protect and improve mental health. Recent studies have shown that logotherapy is an effective method in strengthening positive psychological factors and coping with negative emotions. Logotherapy adopts "Therapy through Meaning" as its basic method. The effectiveness of logotherapy on meaning and hope has been demonstrated in many different samples. No study has been found that focuses on meaning and hope in family members of chronic psychiatric patients. This study aims to determine the effect of a logotherapy-focused psychoeducation program on the meaning in life, hope, and depression levels in families of schizophrenia patients. The results of this study are applicable to family members of individuals diagnosed with schizophrenia. Research hypotheses: H1a: Logotherapy-based psychoeducation applied to family members of individuals diagnosed with schizophrenia will cause an increase in the members' finding and searching for meaning in life, future, positive readiness and expectation, and relationships with themselves and their surroundings subscale scores. H1b: Logotherapy-based psychoeducation applied to family members of individuals diagnosed with schizophrenia will cause a decrease in the members' depression levels.

DETAILED DESCRIPTION:
The resources that will strengthen the family members who play a key role in the treatment of schizophrenia should also be activated. One of these resources that enable people to cope with the difficult events they experience is finding meaning in life. The meaning of life is a basic source of motivation for an individual to live despite everything. In this respect, meaning is a source that helps them maintain their mental balance. Another concept that is considered important in terms of protecting and strengthening the mental health of family members is hope. Hope is defined as setting a goal and taking action to achieve it, and looking for different ways when faced with difficulties. Hope gives caregivers the belief that they can cope with stressful experiences. Therefore, it is important to develop hope in family members of individuals with mental disorders. Today, different therapy methods are applied to protect and improve mental health. Recent studies have shown that logotherapy is an effective method in strengthening positive psychological factors and coping with negative emotions. Logotherapy adopts "Therapy through Meaning" as its basic method. The effectiveness of logotherapy on meaning and hope has been demonstrated in many different samples. No study has been found that focuses on meaning and hope in family members of chronic psychiatric patients. This study aims to determine the effect of a logotherapy-focused psychoeducation program on the meaning in life, hope, and depression levels in families of schizophrenia patients. The results of this study are applicable to family members of individuals diagnosed with schizophrenia. Research hypotheses: H1a: Logotherapy-based psychoeducation applied to family members of individuals diagnosed with schizophrenia will cause an increase in the members' finding and searching for meaning in life, future, positive readiness and expectation, and relationships with themselves and their surroundings subscale scores. H1b: Logotherapy-based psychoeducation applied to family members of individuals diagnosed with schizophrenia will cause a decrease in the members' depression levels.

Type of Research This research was planned as a mixed design study using quantitative and qualitative approaches together. The quantitative phase of the research consists of a prospective, single-blind, randomized controlled study design using a pre-test-post-test design that aims to reveal the effectiveness of Logotherapy-Based Psychoeducation. The qualitative phase of the study will be applied with a phenomenological approach to clarify the attitude changes of the participants in the experimental group during and after the Logotherapy-Focused Psychoeducation Program.

Place and Time of the Research The research is planned to be conducted at the Istanbul Başakşehir Çam and Sakura City Hospital Mental Health and Hospital between December 2022 and November 2023.

Population, Sample and Sample Characteristics of the Research The population of the research will consist of family members of individuals diagnosed with schizophrenia who are followed up at the Başakşehir Çam and Sakura City Hospital Psychiatry Outpatient Clinic, and the sample will consist of family members who meet the inclusion criteria. After the sample size is calculated, randomization will be performed and the experimental and control groups will be determined.

Data Collection Tools Personal Information Form This form, created by the researcher by scanning the relevant literature, consists of 14 questions aimed at determining the sociodemographic and disease-related characteristics of the individual diagnosed with schizophrenia and his/her family member.

The Meaning of Life Scale The meaning of life scale was developed by Steger and colleagues to determine the meaning people find in life and the meaning they seek. The adaptation study for Turkey was conducted by Akın and Taş. The meaning of life scale consists of 10 items on a 7-point Likert type. The scale consists of two subscales, namely current meaning and sought meaning. The total score on the scale varies between 7 and 70. High scores obtained from the scale indicate that the individual has a high level of meaning in life. The internal consistency reliability coefficients of the scale are .82 for the current meaning subscale and .87 for the sought meaning subscale.

Herth Hope Scale The Herth Hope Scale was developed by Dr. Herth in 1991 to determine the hope levels of individuals and was adapted to Turkish by Aslan and colleagues. The scale is a four-point Likert type and consists of 30 items. The scale consists of the sub-dimensions "Future", "Positive readiness and expectation" and "Relationships between oneself and those around oneself". The total hope score varies between 0-90, and the total score for each sub-scale varies between 0-30. High scores obtained from the scale indicate a high level of hope. In the reliability study of the Turkish form of the scale, the Cronbach alpha coefficient was determined as 0.84.

Beck Depression Inventory II The Beck Depression Inventory was first developed by Aeoron T. Beck in 1961 to determine the risk of depression in individuals and to measure the level and severity of depressive symptoms. The validity and reliability of the BDI for the Turkish society was conducted by Çınarbaş et al. The BDI is a three-point Likert-type scale and consists of 21 items. A total score of 0-63 is obtained from the items, and an increase in the total score indicates an increase in depressive symptoms. The cut-off score for the Turkish society is generally accepted as 17.

Semi-structured qualitative interview form The semi-structured interview form to be used for the qualitative interview will be created by the researcher in line with expert opinion while preparing the psychoeducation program.

Data Collection There will be two groups selected by randomization in the study, experimental and control. The logotherapy-based program prepared in line with literature information and expert opinion will be applied to the family members in the experimental group using the focus group interview method.

YÖÖ, HUÖ and BDE will be applied to the family members at the beginning, end and follow-up of the psychoeducation program. In addition, qualitative data will be collected with the Semi-Structured Interview Form developed by the researcher during the follow-up phase.

Data Analysis The collected quantitative data will be brought together and coded. Then, the coded data will be transferred to the SPSS program database and the data will be separated into parametric and nonparametric groups and analyzed with hypothesis analysis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

  * Volunteering to participate in the study
  * Having a family history of schizophrenia diagnosed according to DSM-5 diagnostic criteria
  * An individual diagnosed with schizophrenia being followed up with this diagnosis for at least one year
  * Being over the age of 18

Exclusion Criteria: Being treated or being treated for a mental disorder

* Having received or being receiving psychotherapy Exclusion criteria from the study
* Not attending at least two of the psychoeducation sessions
* An individual diagnosed with schizophrenia being hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-05-03 (Estimated); Primary Completion 2025-08-03 (Estimated); Study Completion 2025-09-03 (Estimated)

PRIMARY OUTCOMES:
Finding meaning in life scale score | first week and eighth week
  The meaning of life scale was developed by Steger and colleagues (1) to determine the meaning people find in life and the meaning they seek. The adaptation study for Turkey was conducted by Akın and Taş (2). The meaning of life scale consists of 10 items on a 7-point Likert type. The scale consists of two subscales, namely current meaning and sought meaning. The total score on the scale varies between 7 and 70. High scores obtained from the scale indicate that the individual has a high level of meaning in life. The internal consistency reliability coefficients of the scale are .82 for the current meaning subscale and .87 for the sought meaning subscale.
Herth Hope Scale Scores | first week and eighth week
  The Herth Hope Scale (HUÖ) was developed by Dr. Herth in 1991 to determine the hope levels of individuals and was adapted to Turkish by Aslan and colleagues. The scale is a four-point Likert type and consists of 30 items. The scale consists of the sub-dimensions "Future", "Positive readiness and expectation" and "Relationships between oneself and those around oneself". The total hope score varies between 0-90, and the total score for each sub-scale varies between 0-30. High scores obtained from the scale indicate a high level of hope. In the reliability study of the Turkish form of the scale, the Cronbach alpha coefficient was determined as 0.84.
Beck Depression Inventory Scores | first week and eighth week
  The Beck Depression Inventory was first developed by Aeoron T. Beck in 1961 to determine the risk of depression in individuals and to measure the level and severity of depressive symptoms. The validity and reliability of the BDI for the Turkish society was conducted by Çınarbaş et al. The BDI is a three-point Likert-type scale and consists of 21 items. A total score of 0-63 is obtained from the items, and an increase in the total score indicates an increase in depressive symptoms. The cut-off score for the Turkish society is generally accepted as 17.
Results of semi-structured qualitative form | tenth week
  The semi-structured interview form to be used for the qualitative interview will be created by the researcher in line with expert opinion while preparing the psychoeducation program.

OTHER OUTCOMES:
Personal İnformation Form | first week
  This form, created by the researcher by scanning the relevant literature, consists of 14 questions aimed at determining the sociodemographic and disease-related characteristics of the individual diagnosed with schizophrenia and his/her family member.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frankl VE. Logotherapy. Isr Ann Psychiatr Relat Discip. 1967;5(2):142-55. No abstract available. PMID 5247330
- [Background] Eskigulek Y, Kav S. Effect of logotherapy counseling program on chronic sorrow, dignity, and meaning in life of palliative care patients: a randomized controlled trial. Support Care Cancer. 2024 Aug 13;32(9):587. doi: 10.1007/s00520-024-08792-w. PMID 39138762
- [Background] Aydin R, Kabukcuoglu K. The effect of logotherapy-based, nurse-guided meaning attribution conversations on women diagnosed with gynecologic cancer: A Turkish pilot study. Women Health. 2023 Sep 14;63(8):599-614. doi: 10.1080/03630242.2023.2249123. Epub 2023 Aug 29. PMID 37642347
- [Background] Sun FK, Hung CM, Yao Y, Fu CF, Tsai PJ, Chiang CY. The Effects of Logotherapy on Distress, Depression, and Demoralization in Breast Cancer and Gynecological Cancer Patients: A Preliminary Study. Cancer Nurs. 2021 Jan/Feb;44(1):53-61. doi: 10.1097/NCC.0000000000000740. PMID 31469671
- [Background] Applebaum AJ, Buda KL, Schofield E, Farberov M, Teitelbaum ND, Evans K, Cowens-Alvarado R, Cannady RS. Exploring the cancer caregiver's journey through web-based Meaning-Centered Psychotherapy. Psychooncology. 2018 Mar;27(3):847-856. doi: 10.1002/pon.4583. Epub 2017 Dec 19. PMID 29136682
- [Background] Shewchun J, Garside BK, Ballik EA, Kwan CC, Elsherbiny MM, Hogenkamp G, Kazandjian A. Pollution monitoring systems based on resonance absorption measurements of ozone with a "tunable" CO(2) laser: some criteria. Appl Opt. 1976 Feb 1;15(2):340-6. doi: 10.1364/AO.15.000340. PMID 20164973
- [Background] Yang X, Zhang P, Jing S, Cheng Y, Cavaletto A. Logotherapy-Based Interventions for Chinese Family Caregivers of Older Adults with Dementia Through Online Groups: A Mixed-Methods Study. J Gerontol Soc Work. 2024 Oct;67(7):865-880. doi: 10.1080/01634372.2024.2326689. Epub 2024 Mar 10. PMID 38461440